CLINICAL TRIAL: NCT04782492
Title: Morphologic Changes of the Saphenous Vein as Y-composite Graft Based on the Left Internal Thoracic Artery Versus Aortocoronary Conduit for Coronary Artery Bypass Grafting: A Prospective Randomized Controlled Trial
Brief Title: IVUS Study for SV Graft: Y-composite vs Aortocoronary Conduit
Acronym: CONFIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ho Young Hwang (Other)
Responsible Party: Sponsor-Investigator, Ho Young Hwang, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-2101-143-1191
Record Dates: First submitted 2021-03-02; First posted 2021-03-04 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Morphologic Change
Keywords: Coronary artery bypass grafting; Saphenous vein; Intravascular ultrasound
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Intervention Model Description: saphenous vein as Y-composite graft based on the left internal thoracic artery versus aortocoronary conduit
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Y-composite graft (Experimental): The saphenous vein is anastomosed to the middle portion of the left internal thoracic artery as Y-composite fashion. Then, left anterior descending artery, if targeted, is bypassed with left internal thoracic artery. Other native coronary arterial targets are bypassed with saphenous vein graft.
  Interventions: Procedure: graft configuration in coronary artery bypass grafting
- aortocoronary conduit (Active Comparator): The saphenous vein is anastomosed to the ascending aorta as aortocoronary fashion. Then, left anterior descending artery, if targeted, is bypassed with left internal thoracic artery. Other native coronary arterial targets are bypassed with saphenous vein graft.
  Interventions: Procedure: graft configuration in coronary artery bypass grafting

INTERVENTIONS:
Procedure: graft configuration in coronary artery bypass grafting — Saphenous vein could be used as Y-composite graft or aortocoronary conduit during coronary artery bypass grafting

SUMMARY:
Left internal thoracic artery (LITA) has been acknowledged as the first graft of choice for coronary artery bypass grafting (CABG). However, it is still not conclusive which one is the best second graft of choice among right internal thoracic artery, radial artery, right gastroepiploic artery, saphenous vein, and etc., as well as its configuration for CABG.

In our institution, saphenous vein has been primarily used for the second graft and we have harvested it with 'No touch technique'. We have been demonstrated the excellent long-term patency of this 'No touch saphenous vein' in many studies. However, it is still unknown which configuration is the better strategy for the saphenous vein as a Y-composite graft based on the left internal thoracic artery versus an aortocoronary conduit. Thus, we aimed to evaluate morphologic change of saphenous vein graft by 1-year intravascular ultrasound (IVUS) study and angiographic patency results between Y-composite graft and aortocoronary conduit.

DETAILED DESCRIPTION:
The enrolled patient underwent routine sternotomy, and left internal thoracic artery (LITA) and saphenous vein (SV) are harvested. After harvest, the patient is randomized to Y-composite group or aortocoronary group.

For Y-composite group, SV is anastomosed to LITA as Y-composite fashion. Then, LITA is anastomosed to left anterior descending artery. SV is anastomosed to the rest of the target vessels with sequential anastomosis technique (e.g. diagonal branch, obtuse marginal branch, posterolateral branch and posteriori descending artery).

For aortocoronary group, LITA is anastomosed to left anterior descending artery. Then, SV is anastomosed to ascending aorta using proximal anastomosis assist device without clamping the aorta. SV is anastomosed to the rest of the target vessels with sequential anastomosis technique (e.g. diagonal branch, obtuse marginal branch, posterolateral branch and posteriori descending artery).

After completion of anastomoses, residual portion of distal SV is collected for microscopic evaluation and measurement of intima-media thickness.

At the 1-year follow-up, IVUS study, in addition to coronary angiography, is performed to evaluate the morphologic changes and measure intima-media thickness of the saphenous vein graft.

ELIGIBILITY:
Inclusion Criteria:

* A patient who is going to receive coronary artery bypass grafting
* Older than 19 years
* Coronary artery bypass grafting is going to be performed with left internal thoracic artery and saphenous vein graft

Exclusion Criteria:

* Other concomitant procedures (e.g. valve or aorta surgery) is planned
* Patients with severe comorbidities which limit the life expectancy of them below 1 year (e.g. terminal cancer)
* Patients whose left internal thoracic artery or saphenous vein is not available due to the low quality, severe injury, or absence of the graft

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Intima-media thickness (IMT) | at postoperative 1 year
  Intima-media thickness measured by intravascular ultrasound (IVUS)

SECONDARY OUTCOMES:
Lumen diameter (LD) | at postoperative 1 year
  Lumen diameter measured by intravascular ultrasound (IVUS)
Graft patency | at postoperative 1 year
  Graft patency measured by coronary angiography
All cause mortality | at postoperative 1 year
  all deaths from any cause
Cardiac death | at postoperative 1 year
  Any death related to cardiac events, including sudden death during follow-up
Target vessel revascularization | at postoperative 1 year
  The number of patients who received any intervention performed for the previously bypassed target vessel during follow-up
Reintervention | at postoperative 1 year
  The number of patients who received any coronary intervention performed during follow-up due to the coronary artery disease

CONTACTS AND LOCATIONS:
Overall Officials: Ho Young Hwang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because it is not allowed by our Institutional Review Board.

REFERENCES:
- [Derived] Sohn SH, Kang Y, Kim JS, Kang J, Hwang HY. Morphologic changes of the no-touch saphenous vein as Y-composite versus aortocoronary grafts (CONFIG Trial). PLoS One. 2025 May 8;20(5):e0322176. doi: 10.1371/journal.pone.0322176. eCollection 2025. PMID 40338976